CLINICAL TRIAL: NCT01351584
Title: Clinical Registry to Present Treatment and Sequences of Treatments in Routine Practice in Germany
Brief Title: Tumour Registry Breast Cancer
Acronym: TMK
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitskreis Klinische Studien (Other); Arbeitsgemeinschaft fur Internistische Onkologie (Other)
Responsible Party: Sponsor
Other Study IDs: IOM TMK; Tumorregister Mammakarzinom (Other: iOMEDICO AG)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Advanced Breast Cancer; Epidemiology; Registry; Health Services Research; Germany; Palliative Treatment; Adjuvant Drug Therapy; Nutrition Assessment; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The registry aims to collect and analyse information on the antineoplastic treatment of breast cancer in daily routine practice of office-based and clinic-based medical oncologists in Germany.

DETAILED DESCRIPTION:
The TMK is a prospective, longitudinal, nation wide cohort study with the purpose to record information on the antineoplastic treatment of breast cancer in Germany. The registry will follow patients for up to five years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics, biomarker testing and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

The impact of nutrition (MaNut) and physical activity (MaNut) on the course of the adjuvant disease will be examined, as well as long-term effects of adjuvant treatment (MaTox) and the multiple patient-reported outcomes (MaLife).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* 18 years and older
* Antineoplastic or antihormonal treatment

Exclusion Criteria:

* No breast cancer
* Below 18 years
* No antineoplastic or antihormonal treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients undergoing antineoplastic or antihormonal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Course of Antineoplastic Treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Tesch, MD, Study Chair

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fietz T, Tesch H, Rauh J, Boller E, Kruggel L, Janicke M, Marschner N; TMK-Group (Tumour Registry Breast Cancer). Palliative systemic therapy and overall survival of 1,395 patients with advanced breast cancer - Results from the prospective German TMK cohort study. Breast. 2017 Aug;34:122-130. doi: 10.1016/j.breast.2017.05.014. Epub 2017 Jun 3. PMID 28586735
- [Background] Schroder J, Fietz T, Kohler A, Petersen V, Tesch H, Spring L, Fleitz A, Janicke M, Marschner N; TMK-Group (Tumour Registry Breast Cancer). Treatment and pattern of bone metastases in 1094 patients with advanced breast cancer - Results from the prospective German Tumour Registry Breast Cancer cohort study. Eur J Cancer. 2017 Jul;79:139-148. doi: 10.1016/j.ejca.2017.03.031. Epub 2017 May 8. PMID 28494404
- [Background] Hurtz HJ, Tesch H, Gohler T, Hutzschenreuter U, Harde J, Kruggel L, Janicke M, Marschner N; TMK-Group (Tumour Registry Breast Cancer). Persistent impairments 3 years after (neo)adjuvant chemotherapy for breast cancer: results from the MaTox project. Breast Cancer Res Treat. 2017 Oct;165(3):721-731. doi: 10.1007/s10549-017-4365-7. Epub 2017 Jul 5. PMID 28677012
- [Background] Fietz T, Zahn MO, Kohler A, Engel E, Frank M, Kruggel L, Janicke M, Marschner N; TMK-Group (Tumour Registry Breast Cancer). Routine treatment and outcome of breast cancer in younger versus elderly patients: results from the SENORA project of the prospective German TMK cohort study. Breast Cancer Res Treat. 2018 Jan;167(2):567-578. doi: 10.1007/s10549-017-4534-8. Epub 2017 Oct 13. PMID 29030786
- [Background] Dorfel S, Steffens CC, Meyer D, Tesch H, Kruggel L, Frank M, Janicke M, Marschner N; TMK-Group (Tumour Registry Breast Cancer). Adjuvant chemotherapeutic treatment of 1650 patients with early breast cancer in routine care in Germany: data from the prospective TMK cohort study. Breast Cancer. 2018 May;25(3):275-283. doi: 10.1007/s12282-017-0823-7. Epub 2017 Dec 4. PMID 29204847
- [Background] Marschner N, Trarbach T, Rauh J, Meyer D, Muller-Hagen S, Harde J, Dille S, Kruggel L, Janicke M; TMK-Group (Tumour Registry Breast Cancer). Quality of life in pre- and postmenopausal patients with early breast cancer: a comprehensive analysis from the prospective MaLife project. Breast Cancer Res Treat. 2019 Jun;175(3):701-712. doi: 10.1007/s10549-019-05197-w. Epub 2019 Mar 13. PMID 30868393